CLINICAL TRIAL: NCT03250026
Title: Cooperation for Patients With Common Mental Disorders: Care Manager Function at the Primary Care Centre and Intervention at the Workplace - CO-WORK-CARE
Brief Title: Cooperation for Primary Care Patients on Sick Leave for CMD: Care Manager and Workplace Intervention - CO-WORK-CARE
Acronym: CO-WORK-CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 459-17
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder; Anxiety Disorders
Keywords: primary care; convergence dialogue; sick leave; care manager
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Case Managers

STUDY DESIGN:
Intervention Model Description: Pragmatic randomised controlled trial; randomisation on primary care centre level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Workplace dialogue) (Experimental): Intervention: Work place convergence dialogue contact
  Interventions: Behavioral: Workplace convergence dialogue; Behavioral: Care Manager
- Care Manager (Active Comparator): Intervention: Care Manager contact 12 weeks (Care as usual)
  Interventions: Behavioral: Care Manager

INTERVENTIONS:
Behavioral: Workplace convergence dialogue — Work place contact as a convergence dialogue between the employer and employee with the Rehab Coordinator as a guide
  Arms: Intervention (Workplace dialogue)
Behavioral: Care Manager — Regular contact Care Manager during around 12 weeks

SUMMARY:
This study aims to evaluate whether a convergence dialogue during sick leave, between the employee and the employer, with the Primary Care Centre Rehab Coordinator as discussion leader, leads to reduced sick leave time compared to those individuals who only have contact with a Care Manager during the period of sick leave. The study will be performed as a randomised controlled trial with randomisation at the PCC level where intervention PCCs offers a convergence dialogue meeting with the work place representative during sick leave in addition to Care Manager contact.

DETAILED DESCRIPTION:
In Sweden sick leave time and frequency are increasing. This is primarily in the area of common mental disorders (CMD), and CMD is now the most common single cause of sickness absence. Primary care is the area in which most individuals with mental illness seek care and also receive care. A Care Manager function at the primary care centre (PCC) where the Care Manager is responsible for the support and close contact with patients with CMD and act as the "spider in the web" and combine patient support with other measures, have been shown to have beneficial effects for depression course. In Region Västra Götaland an implementation of the Care Manager function at the PCC has been set out, and the function is now available in nearly 100 PCCs in the region. The present study aims to evaluate whether a convergence dialogue during sick leave, between the employee and the employer, with the PCCs Rehab Coordinator as discussion leader, leads to reduced sick leave time compared to those individuals who only have contact with the Care Manager during the period of sick leave. The study will be performed as pragmatic randomised controlled trial with randomisation at the PCC level. Around 20 PCCs with a Care Manager function for patients on sick-leave with CMD diagnosis will be recruited and randomized to intervention where patients in addition to a Care Manager contact (12 weeks) will have one convergence dialogue meeting with the work place representative during sick leave. Control PCCs will give Care Manager contact 12 weeks only.

ELIGIBILITY:
Inclusion Criteria:

Patients attending primary care centers with care manager function

* aged >=18 to 67 years
* diagnosed with a new (< 1 month) depression diagnose (F32, F33), anxiety syndrome (F41, F48) or stress related adjustment disorder (F43)
* on sick-leave > 14 days

Exclusion Criteria:

* Bipolar disorder
* psychosis
* addiction
* other serious mental disorder
* suicidal ideation or earlier suicide attempt
* cognitive impairment or not speaking/understanding Swedish

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Net and gross sick-leave days | 12 months
  number of net and gross sick-leave days during 12 months

SECONDARY OUTCOMES:
Depressive symptoms | 6 and 12 months
  Change of depressive symptoms Montgomery-Asberg Depression Rating Scale - Self rating version (MADRS-S) Range 0-60 (Total score) Low score better outcome
Anxiety symptoms | 6 and 12 months
  Change of anxiety symptoms Generalized Anxiety Disorder 7-item (GAD-7) scale Range 0-15 (total score) low score better outcome
Quality-of-life questionnaire score | 6 and 12 months
  Change of quality of life EuroQoL-5 Dimension Questionnaire(EQ-5D) Range 0-1.0(total score) low score worst outcome
Work ability | 6 and 12 months
  Change of work ability Work Ability Index (WAI) Range 7-49 (total score) low score worst outcome
Exhaustion | 6 and 12 months
  Change of Exhaustion Karolinska Exhaustion Disorder Scale (KEDS) Range 0-54 (total score) low score better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Björkelund, prof, Principal Investigator — Göteborg University
Locations (1):
- Department of Primary Health Care, Sahlgrenska Academy, Gothenburg, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participants will be made available to other researchers, provided reasonable request by personal contact, as soon as publication of results is effected.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available after 12 months after study completion/ alternatively as soon as publication of results is effected.
Access Criteria: Data access will be reviewed by an external independent review panel.

REFERENCES:
- [Background] Petersson EL, Tornbom K, Hange D, Nejati S, Jerlock M, Wikberg C, Bjorkelund C, Svenningsson I. The experiences of care managers and rehabilitation coordinators of a primary care intervention to promote return to work for patients with common mental disorders: a qualitative study. BMC Fam Pract. 2020 Dec 18;21(1):272. doi: 10.1186/s12875-020-01348-x. PMID 33339512
- [Background] Petersson EL, Tornbom K, Bjorkelund C, Jerlock M, Hange D, Udo C, Svenningsson I. Process evaluation of the CO-WORK-CARE model: Collaboration and a person-centred dialogue meeting for patients with common mental disorder in primary health care. Scand J Caring Sci. 2024 Sep;38(3):602-613. doi: 10.1111/scs.13268. Epub 2024 May 8. PMID 38718100
- [Background] Saxvik A, Svenningsson I, Tornbom K, Petersson EL, Bjorkelund C, Gabartaite G, Hange D. GPs' experiences of a collaborative care model for patients with common mental disorders who need sick leave certification: a qualitative study. BJGP Open. 2022 Dec 20;6(4):BJGPO.2022.0042. doi: 10.3399/BJGPO.2022.0042. Print 2022 Dec. PMID 35977733
- [Background] Saxvik A, Tornbom K, Petersson EL, Hange D, Nejati S, Bjorkelund C, Svenningsson I. Experiences of patients with common mental disorders concerning team-based primary care and a person-centered dialogue meeting: An intervention to promote return to work. PLoS One. 2022 Jul 8;17(7):e0271180. doi: 10.1371/journal.pone.0271180. eCollection 2022. PMID 35802679
- [Background] Bjorkelund C, Petersson EL, Svenningsson I, Saxvik A, Wiegner L, Hensing G, Jonsdottir IH, Larsson M, Wikberg C, Ariai N, Nejati S, Hange D. Effects of adding early cooperation and a work-place dialogue meeting to primary care management for sick-listed patients with stress-related disorders: CO-WORK-CARE-Stress - a pragmatic cluster randomised controlled trial. Scand J Prim Health Care. 2024 Sep;42(3):378-392. doi: 10.1080/02813432.2024.2329212. Epub 2024 Mar 31. PMID 38555865
- [Result] Bjorkelund C, Saxvik A, Svenningsson I, Petersson EL, Wiegner L, Larsson M, Tornbom K, Wikberg C, Ariai N, Nejati S, Hensing G, Hange D. Rehabilitation cooperation and person-centred dialogue meeting for patients sick-listed for common mental disorders: 12 months follow-up of sick leave days, symptoms of depression, anxiety, stress and work ability - a pragmatic cluster randomised controlled trial from the CO-WORK-CARE project. BMJ Open. 2023 Jun 9;13(6):e074137. doi: 10.1136/bmjopen-2023-074137. PMID 37295824
- [Result] Svenningsson I, Bjorkelund C, Hange D, Wiegner L, Ariai N, Petersson EL. Symptom patterns in patients newly sick listed for common mental disorders and associations with work-related and socioeconomic factors: a cross-sectional study in Swedish primary care. BMJ Open. 2022 Jul 8;12(7):e054250. doi: 10.1136/bmjopen-2021-054250. PMID 35803640